CLINICAL TRIAL: NCT07397767
Title: Development of Quantitative Parameter of Upper Extremity Function in Patients With Brain Disorder Using Smart-Board and Smart-Glove, Single-Center, Prospective Study
Brief Title: Development of Quantitative Parameter of Upper Extremity Function in Patients With Brain Disorder Using Smart-Board and Smart-Glove.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Hyuk Chang, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-11-105; RS-2023-00248118 (Other Grant/Funding Number: Korea Medical Device Development Fund)
Record Dates: First submitted 2026-01-20; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Brain Disorder; Smart Device Rehabilitation
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smart Device User (Experimental): Smart Device User
  Interventions: Device: smart device

INTERVENTIONS:
Device: smart device — Participants will undergo two sessions of upper-limb movement assessment using the smart board and smart glove on the day of the clinical trial. Simultaneously, video recordings will be obtained using a mobile camera. These procedures will be used to collect quantitative data on upper-limb movements.

SUMMARY:
The aim of this study is to develop a novel quantitative metric for assessing upper-limb function in patients with neurological disorders. This will be accomplished by analyzing performance data obtained from a smart board and smart glove system and comparing these data with conventional clinical assessment methods currently used to evaluate upper-limb impairment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older.
* Patients with upper-limb functional impairment due to neurological conditions such as stroke, cerebral palsy, brain tumor, traumatic brain injury, or Parkinson's disease.

Exclusion Criteria:

* Patients with progressive neurological disorders or those in a state of hemodynamic instability.
* Patients with severe cognitive impairment (MMSE < 10) or significant communication difficulty due to language disorders.
* Any other condition in which the investigator determines that participation in the study is inappropriate.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
validity | the day of the study procedures
  To examine the correlation between the primary outcome measure (FM-UE) and the trunk rehabilitation assessment model derived from mobile camera, smart board, and smart glove data.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea